CLINICAL TRIAL: NCT02464462
Title: The Role of Vitamin D and Calcium Supplementation in the Pathogenesis of Type 2 Diabetes Mellitus
Brief Title: The Role of Vitamin D3 and Calcium Supplementation in Attenuating T2DM Severity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: York University (Other)
Collaborators: Women's Health in Women's Hands Community Health Center (Unknown)
Responsible Party: Principal Investigator, MAZEN J HAMADEH, Associate Progessor, York University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 220; STU 2013-024 (Other: York University Research Ethics Board)
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: serum calcidiol; T2DM; vitamin D3 supplementation; post-menopausal women; ethnic diverse; calcium supplementation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- CaD Group (Experimental): This arm received total of 1800 IU of vitamin D3 and 720 mg of calcium
  Interventions: Dietary Supplement: vitamin D3 and calcium
- Placebo Group (Placebo Comparator): This arm received rice powder pills
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D3 and calcium — 1800 IU vitamin D3 plus 720 mg Calcium
  Arms: CaD Group
Other: Placebo — Rice powder pills
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to investigate the effect of vitamin D3 and calcium supplementation in attenuating type 2 diabetes mellitus outcomes in ethnic diverse, diabetic patiens.

DETAILED DESCRIPTION:
Subjects of this study received a total of 1800 IU vitamin D3 and 720 mg of calcium per day for 3 years. The study was conducted in Toronto, Ontario, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Non-white, post menopausal female
* Have access to Community Health Center

Exclusion Criteria:

* neurodegenerative disease
* kideny disease
* gluten allergy

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Serum calcidiol | 3 years

SECONDARY OUTCOMES:
Fasting insulin | 3 years
Parathyroid Hormone | 3 years
Fasting blood glucose | 3 years
Glycated Hemoglobin | 3 years